CLINICAL TRIAL: NCT06489717
Title: Comparative Study of Sleep Disordered Breathing (SDB) in Patients With High Altitude Pulmonary Hypertension Permanently Residing Above 2500 Meters When Assessed Near Resident High Altitude (HA) at 3200 m vs. at Low Altitude (LA) 760 m
Brief Title: High Altitude Residents With High Altitude Pulmonary Hypertension (HAPH), SDB Assessed at HA (3200 m) vs LA (760 m)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HAPH_HAvsLA_SDB
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; High Altitude; Sleep disordered breathing
MeSH Terms: conditions — Pulmonary edema of mountaineers; Hypertension, Pulmonary; Hypoxia; Altitude Sickness; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Each highlander with HAPH will be assessed for SDB at 3200 m and at 760 m according to a prospective study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessments at 3200 m and 760 m, respectively (Experimental): Participants will have a SDB assessment near their resident altitude at 3200 m and after relocation to 760 m after 1 and 7 days
  Interventions: Other: SDB assessment

INTERVENTIONS:
Other: SDB assessment — SDB will be assessed by respiratory polygraphy according to clinical standards

SUMMARY:
To study the effect of relocation from 3200m (Aksay) to 760m (Bishkek) in highlanders with High Altitude Pulmonary Hypertension (HAPH) who permanently live >2500m on sleep disordered breathing

DETAILED DESCRIPTION:
This research in highlanders with HAPH diagnosed by echocardiography and defined by a RV/RA >30 mmHg who permanently live at HA >2500 m will have nocturnal respiratory sleep studies near their living altitude in Aksay at 3200 m and on night 1 and 6 at 760m after relocation.

ELIGIBILITY:
Inclusion Criteria:

* Permanently living >2500 m
* HAPH diagnosed with a minimum RV/RA of 30 mmHg assessed by echocardiography at an altitude of 3200 m
* Written informed consent

Exclusion Criteria:

* Highlanders who cannot follow the study investigations,
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, heavy smoking >20 cigarettes/day or >20 pack-years.
* Coexistent unstable systemic hypertension or coronary artery disease that required adjustment of medication within the last 2 months
* Regular use of medication that affects control of breathing (benzodiazepines, opioids, acetazolamide)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Mean nocturnal SpO2 during the first night at LA vs HA | night 1 at 760 m compared to 3200 m.
  Change in mean nocturnal SpO2 (%) between LA (760 m) vs HA (3200 m)

SECONDARY OUTCOMES:
Mean nocturnal SpO2 during the sixth night at LA vs HA | night 6 at 760 m compared to 3200 m.
  Change in mean nocturnal SpO2 (%) between LA (760 m) vs HA (3200 m)
Time spent with SpO2<90% at LA vs HA | night 1 and night 6 at 760 m compared to 3200 m.
  Change in time spent with SpO2<90% between LA (760 m) vs HA (3200 m)
AHI at LA vs HA | night 1 and night 6 at 760 m compared to 3200 m.
  Change in apnea-hypopnea index (AHI) between LA (760 m) vs HA (3200 m)
ODI at LA vs. HA | night 1 and night 6 at 760 m compared to 3200 m.
  Change in oxygen desaturation index (ODI) between LA (760 m) vs HA (3200 m)
Time spent with periodic breathing at LA vs. HA | night 1 and night 6 at 760 m compared to 3200 m.
  Change in time spent with periodic breathingbetween LA (760 m) vs HA (3200 m)
Heart rate variability at LA vs. HA | night 1 and night 6 at 760 m compared to 3200 m.
  Change in heart rate variability between LA (760 m) vs HA (3200 m)
ECG markers of repolarization at LA vs. HA | night 1 and night 6 at 760 m compared to 3200 m.
  Change in electrocardiogram (ECG) markers of repolarization (QT time) between LA (760 m) vs HA (3200 m)
pulse transit time drops at LA vs. HA | night 1 and night 6 at 760 m compared to 3200 m.
  Change in pulse transit time drops between LA (760 m) vs HA (3200 m)

CONTACTS AND LOCATIONS:
Overall Officials: Talant M Sooronbaev, Prof. Dr., Principal Investigator — National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov; Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- Aksay Medical Center, Aksay Plateau, Naryn, Kyrgyzstan, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided